CLINICAL TRIAL: NCT07307417
Title: Functional Respiratory Tract Dysfunctions in Individuals With Obesity Undergoing Experimental Inspiratory Muscle Training.
Brief Title: Assessment of Respiratory Dysfunction in Obesity and the Use of IMT.
Acronym: IMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Paulina Okrzymowska, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 00913
Record Dates: First submitted 2025-11-26; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight; Inflammation; Ventilation Disorders
Keywords: inspiratory muscle training; obesity; ventilation disorders; inflammation; forced oscillation technique; spirometry
MeSH Terms: conditions — Obesity; Overweight; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMT Group (Experimental)
  Interventions: Device: inspiratory muscle training
- placebo-IMT (Placebo Comparator)
  Interventions: Device: placebo-IMT
- Control group (No Intervention): No Intervention: IMT Control Group - IMT Control Group - participants who will not complete the IMT cycle.

INTERVENTIONS:
Device: inspiratory muscle training — The IMT experimental group will undergo training with a load of 30% of PImax, assessed in the first inspiratory muscle strength test. Training will be conducted twice a day, with 30 breaths in each training session. From the second week onwards, the training load will be increased by 10% each week. The maximum load will be 60% of PImax. The intervention will last 6 weeks and will be performed daily.
  Arms: IMT Group
Device: placebo-IMT — The control group will perform simulated inspiratory muscle training with a constant load of 15% PImax. Training will take place 7 times a week, 60 breaths once a day. The intervention will last 6 weeks and will be performed daily.
  Arms: placebo-IMT

SUMMARY:
The aim of the project will be to assess the functional condition of the respiratory tract and inflammation resulting from obesity, as well as the possibility of using inspiratory muscle training as a factor reducing the occurrence of dysfunction in the respiratory system.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed obesity, BMI equal to or greater than 30 kg/m2
* age between 30 and 60 (women and men),
* consent of the subject.

Exclusion Criteria:

* respiratory diseases requiring pharmacological treatment,
* acute illness that may affect the training programme: e.g. infection, renal failure,
* mental impairment preventing cooperation,
* mental disorders preventing contact and cooperation with the patient,
* pacemaker,
* pregnancy
* implanted electronic
* medical implants
* epilepsy
* metal implants.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | Baseline and after 6 weeks (post-intervention)
  Respiratory function testing (spirometry) will be performed in accordance with the guidelines of the American Thoracic Society and the European Respiratory Society. The respiratory function test will include the following parameters: forced vital capacity (FVC)[FVC in liters], forced expiratory volume in one second (FEV1) [FEV1 in liters], peak expiratory flow (PEF)[PEF in liters/second], vital capacity (VC) [VC in liters], maximum expiratory flow at 25%, 50% and 75% FVC (MEF 25-75%) [MEF 25-75% in liters], maximal inspiratory flow (MIF50) [MIF in liters], maximal expiratory Flow at 50% of vital capacity (MEF50) and maximal inspiratory flow at 50% of vital capacity (MIF50) (MEF50/MIF50) [MEF50/MIF50 in liters].
Respiratory muscle strength (PImax/PEmax) | Baseline and after 6 weeks (post-intervention)
  Respiratory Muscle Strength (PImax/PEmax) by assessing maximum inspiratory pressure (PImax in kilopascal,kPa) and expiratory pressure (PEmax in kilopascal,kPa).
  This measurement is to evaluate the potential effect of the intervention on the strength of inspiratory and expiratory muscles, particularly the potential to improve respiratory muscle performance and enhance overall ventilatory capacity in individuals with reduced respiratory muscle strength.
Forced oscillation technique (FOT) | Baseline and after 6 weeks (post-intervention)
  respiratory mechanics parameter: resistance (Rrs)[Rrs in kPa·s·L-¹], reactance (Xrs) [Xrs in kPa·s·L-¹], resonant Frequency (Fres): The frequency where Xrs = 0 (reactance cancels out).
  This measurement is to evaluate the potential effect of the intervention on airway resistance and reactance, particularly the potential to improve lung mechanics and detect subtle changes in airway function in individuals with impaired or fluctuating respiratory function.
Laboratory tests | Baseline and after 6 weeks (post-intervention)
  inflammatory cytokine profile and CRP (IL-1β, IL-6, IL-8, IL-10, IL-12, TNF-α, CRP), lipid profile.
  Systemic inflammation parameter and lipid profile, this measurement is to evaluate the potential effect of the intervention on inflammatory status, particularly the potential to modify circulating cytokine levels and acute-phase response markers. Laboratory analyses will be performed by qualified diagnostic personnel. Blood samples will be collected into plasma separator tubes (containing lithium-heparin gel), centrifuged, and analyzed. The following parameters will be used for the assessment: interlukin-1β, interlukin-6, interlukin-8, interlukin-10, interlukin-12, tumor necrosis factor-alpha (TNF-α), C-reactive protein (CRP), lipid profile (HDL, LDL, TG). The study will be performed once in all study participants and a second time in those undergoing inspiratory muscle training to assess changes in systemic inflammation associated with the intervention.

SECONDARY OUTCOMES:
Body Composition (Bioelectrical Impedance Analysis, BIA) | Baseline and after 6 weeks (post-intervention)
  Body composition parameter - this measurement assesses: Total Body Water (TBW) [TBW in Liters], Fat-Free Mass (FFM) [FFM in Kilograms], Fat Mass (FM) [FM in Kilograms], Body Fat Percentage (%) in Percentage (%), Height (H) [H in Centimeters], Weight (BW) [BW in Kilograms].
World Health Organization - Quality of Life - BREF (WHOQOL-BREF) | Baseline and after 6 weeks (post-intervention)
  Quality of life parameter - WHOQOL-BREF. This measurement aims to assess participants' perceptions of their quality of life in the physical, mental, social, and environmental areas, in particular the potential to improve the overall well-being and daily functioning of individuals undergoing intervention. The numerical score in each domain reflects individual perceptions of quality of life. Scores are determined on a five-point scale, with a possible range of 4 to 20 points in each domain. The higher the score, the higher the quality of life.
International Physical Activity Questionnaire - short version (IPAQ - short version) | Baseline and after 6 weeks (post-intervention)
  Physical activity parameter. This measure aims to assess participants' physical activity levels, specifically the potential to increase overall activity, reduce sedentary behavior, and monitor changes in daily movement patterns in individuals undergoing the intervention. In IPAQ-SF, physical activity level is measured in MET units (MET - Metabolic Equivalent of Task) [MET - min/week]. High physical activity level is >3000 MET-min/week, moderate is 600-3000 MET-min/week, and low is <600 MET-min/week.

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Kałka, prof., Principal Investigator — Wroclaw University of Health and Sport Sciences; Krystyna Rożek-Piechura, prof., Study Director — Wroclaw University of Health and Sport Sciences; Paulina Okrzymowska, Principal Investigator — Wroclaw University of Health and Sport Sciences
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Dolny Śląsk, Poland

IPD SHARING:
Plan to Share IPD: No